CLINICAL TRIAL: NCT03790748
Title: Comparison of Dural Puncture Epidural Technique Versus Conventional Epidural Technique for Adequate Anesthesia During Vaginal Surgeries
Brief Title: Regional Blocks of Gynecological Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Ali Abdelhaleem Abdelrahman, Lecturer of Anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IUD2900
Record Dates: First submitted 2018-12-23; First posted 2019-01-02 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Gynecologic Disease Requiring Vaginal Operation Under Neuraxial Anesthesia
Keywords: Neuraxial Technique, Epidural Technique, Dural Puncture Epidural Technique, Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Epidural Technique (Experimental): Procedure: Standard Lumbar Epidural Block using Touhy Epidural Needle (18G) at L4-5 inter-space and Epidural Catheter (20G) was inserted then bupivacaine 0.5% 15-20 ml with 50ug fentanyl was given.
  Interventions: Procedure: 25G Dural Puncture Epidural Technique; Procedure: 27G Dural Puncture Epidural Technique
- Dural Puncture Epidural Technique using pencil-point 25G Whitacre needle (Active Comparator): Procedure: 25G Dural Puncture Epidural Block at L4-5 inter-space then bupivacaine 0.5% 15-20 ml with 50ug fentanyl was given.
  Interventions: Procedure: Standard Lumbar Epidural Technique; Procedure: 27G Dural Puncture Epidural Technique
- Dural Puncture Epidural Technique using pencil-point 27G Whitacre needle (Active Comparator): Procedure: 27G Dural Puncture Epidural Block at L4-5 inter-space then bupivacaine 0.5% 15-20 ml with 50ug fentanyl was given.
  Interventions: Procedure: Standard Lumbar Epidural Technique; Procedure: 25G Dural Puncture Epidural Technique

INTERVENTIONS:
Procedure: Standard Lumbar Epidural Technique — Standard Lumbar Epidural Technique at L4-5 inter-space using 0.5%Bupivacaine and Fentanyl.
  Arms: Dural Puncture Epidural Technique using pencil-point 25G Whitacre needle; Dural Puncture Epidural Technique using pencil-point 27G Whitacre needle
Procedure: 25G Dural Puncture Epidural Technique — 25G Dural Puncture Epidural Technique at L4-5 inter-space using 0.5%Bupivacaine and Fentanyl.
  Arms: Conventional Epidural Technique; Dural Puncture Epidural Technique using pencil-point 27G Whitacre needle
Procedure: 27G Dural Puncture Epidural Technique — 27G Dural Puncture Epidural Technique at L4-5 inter-space using 0.5%Bupivacaine and Fentanyl.
  Arms: Conventional Epidural Technique; Dural Puncture Epidural Technique using pencil-point 25G Whitacre needle

SUMMARY:
This study will be conducted on 273 patients of ASA grade I and II aged from 25 to 55 years and presented for elective vaginal surgeries such as vaginal hysterectomy, repair of prolapse Patients will be divided into three equal groups; group A control group for conventional epidural technique(n=91), group B for dural puncture epidural with 27G pencil point Whitacre spinal needle (n=91) and group C for dural puncture epidural with 25G pencil point Whitacre spinal needle(n=91). Randomization will be done using computer generated number and concealed using sequentially numbered sealed opaque envelope.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* Height(150-170 cm)

Exclusion Criteria:

* patient refusal
* hypersensitivity to local anesthetic drugs
* bleeding disorders and coagulopathy(platelets count less than 80000,INR less than 1.5 or therapeutic dose of anticoagulant).

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 273 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
incidence of bilateral sacral blockade | Up to 30 minutes after local anesthetic injection
  Sensory blockade was evaluated using a non-traumatic pinprick stimulus starting at the S2 dermatome and moving in a caudad direction (measured every 2 minutes)

SECONDARY OUTCOMES:
Onset of sensory blockade | Up to 30 minutes after local anesthetic injection
Maximum achieved sensory level | Up to 30 minutes after local anesthetic injection
Time to achieve the maximum sensory level | Up to 30 minutes after local anesthetic injection
Onset of motor blockade | Up to 30 minutes after local anesthetic injection
Time to complete motor block | Up to 30 minutes after local anesthetic injection
Duration of sensory block | Assessed every 20 minutes after achieving highest dermatome level of sensory analgesia
  Time to two segmental dermatomes regression
Duration of motor block | Assessed every 20 minutes after achieving Bromage 3 motor block
  Time interval from achievement of Bromage 1 to regression of motor blockade to Bromage 1
Duration of analgesia | Time for requirement for rescue analgesia or VAS pain score >3 as postoperatively
  Time from onset of sensory block to first complain of pain postoperatively as the epidural catheter will be removed after the surgery finished
Number of epidural top-ups | Number of extra doses of local anesthetic given after injection of local anesthetic loading dose till end of the surgery
Sedation score | Assessed every 20 minutes during the surgical procedure and postoperatively
Hemodynamic parameters | Assessed every 5 minutes from the start of anesthetic procedures till transfer the patients to the rooms
Perioperative side effects | During surgical period up to 7 days post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Reham Ali Abdelrahman, M.D., Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Department of Anesthesia, Surgical ICU, and Pain Management, Cairo
  - Reham Ali Abdelrahman, Cairo